CLINICAL TRIAL: NCT03837990
Title: Development of Prediction Model of Treatment Outcome of Helicobacter Pylori Eradication Through "One Sequencing Find All" Approach: With Whole Exome Sequencing for Host and Target Sequencing for Bacteria at Once
Brief Title: One Sequencing Find All for Helicobacter Pylori Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20181011/20-2018-80/112
Record Dates: First submitted 2019-02-11; First posted 2019-02-12 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-02

CONDITIONS: Helicobacter Pylori Infection; Resistant Infection
Keywords: Whole genome sequencing; Polymorphism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gastric mucosal tissue sample will be used by remnant tissue of CLO test during gastroduodenoscopy. To protect information of participants, we plan to encrypt/anonymize all identifiers of the subjects and store them in a separate database. Whole genome data will be stored in the database of the laboratory of Seoul National University Hospital, and the patient's medical record information (EMR data) will be stored separately.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Helicobacter Pylori eradication therapy — Eradication therapy includes the administration of a proton pump inhibitor (PPI) and antibiotics. Triple therapy with a PPI (lansoprazole or esomeprazole), clarithromycin, and amoxicillin is the first-line regimen. Quadruple therapy with a PPI, bismuth, metronidazole, and tetracyclin is the second-line therapy.
  Other Names: next-generation sequencing of HP strain and host

SUMMARY:
The aim of this study is to Identify antibiotic resistance gene mutations in Helicobacter pylori (HP) and genetic diversity of drug metabolism for antibiotics and proton pump inhibitors (PPIs) in patients with HP infection using next-generation sequencing (NGS). The mutation of host/HP strain will be investigated by single NGS, and the eradication results according to genetic polymorphism of host/HP strain will be analyzed.

DETAILED DESCRIPTION:
This study is a prospective observational study for the Helicobacter pylori (HP) infected patients on typical gastroduodenoscopy (EGD) at Boramae Hospital, Seoul, Korea.

The presence of antibiotic resistance genes of HP and the diversity of the pharmacokinetic genotypes of the subjects will be investigated by performing single next-generation sequencing (NGS) analysis using gastric mucosal tissue samples of the HP infected subjects.

The purpose of this study is to collect data on the antimicrobial resistance mutation of HP (23S rRNA gene, pbp1 gene, rdxA, frxA, frxB gene, 16S rRNA, gyrA, gyrB gene, and Cag A gene) and to investigate the genetic diversity on the metabolism of antibiotics and proton pump inhibitors (CYP enzyme) in a Korean population.

The investigators are going to compare the results of standard eradication therapy according to the resistance mutation of HP and drug genetic diversity of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* CLO test positive
* Findings of gastric ulcer, atrophic gastritis on gastroduodenoscopy
* Agreed to HP eradication therapy and accept to follow-up
* Agreed to participating in the study

Exclusion Criteria:

* History of previous HP eradication treatment
* History of partial gastrectomy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: H. pylori-positive healthy patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Eradication rate of HP infection | 12 months
  intent to treat and per protocol analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ju Han Kim, MD, Study Director — Division of Biomedical Informatics,Seoul National University College of Medicine
Locations (1):
- Seoul National University Boramae Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Graham DY, Fischbach L. Helicobacter pylori treatment in the era of increasing antibiotic resistance. Gut. 2010 Aug;59(8):1143-53. doi: 10.1136/gut.2009.192757. Epub 2010 Jun 4. PMID 20525969
- [Background] Sugimoto M, Furuta T. Efficacy of tailored Helicobacter pylori eradication therapy based on antibiotic susceptibility and CYP2C19 genotype. World J Gastroenterol. 2014 Jun 7;20(21):6400-11. doi: 10.3748/wjg.v20.i21.6400. PMID 24914361
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Gisbert JP, Kuipers EJ, Axon AT, Bazzoli F, Gasbarrini A, Atherton J, Graham DY, Hunt R, Moayyedi P, Rokkas T, Rugge M, Selgrad M, Suerbaum S, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study Group and Consensus panel. Management of Helicobacter pylori infection-the Maastricht V/Florence Consensus Report. Gut. 2017 Jan;66(1):6-30. doi: 10.1136/gutjnl-2016-312288. Epub 2016 Oct 5. PMID 27707777